CLINICAL TRIAL: NCT01538420
Title: Assessment of the Muscle Protein Fractional Synthesis Rate Induced by Repeated Administrations of GLPG0492 to Healthy Male Subjects and Assessment of the Safety, Tolerability and Pharmacokinetics of Repeated Administrations of GLPG0492 to Healthy Postmenopausal Women.
Brief Title: GLPG0492 Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0492-CL-103; 2011-004743-41 (EudraCT Number)
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — 4-(4-(hydroxymethyl)-3-methyl-2,5-dioxo-4-phenylimidazolidin-1-yl)-2-(trifluoromethyl)benzonitrile

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0492 oral solution (Experimental): Multiple ascending doses once daily for 7 days (part 1) or 14 days (part 2), starting at 0.5 mg/day
  Interventions: Drug: GLPG0492
- Placebo (Placebo Comparator): Placebo oral solution, once daily for 7 days (part 1) or 14 days (part 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0492 — Oral solution
  Arms: GLPG0492 oral solution
Drug: Placebo — Placebo oral solution
  Arms: Placebo

SUMMARY:
GLPG0492 is a selective androgen receptor modulator: the compound should help protect against (or help restore) muscle loss in case of immobilization (e.g. after orthopedic surgery) or due to aging (androgenic effect), but without anabolic effects (e.g. effect on testosterone). In the first part of the current study it will be tested whether GLPG0492 given orally to healthy male volunteers increases the protein synthesis in muscle, as measured by the uptake into the muscle of intravenously infused phenylalanine.

In the second part of the study, the effect of the compound on the "hormone household" in healthy, postmenopausal women will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years (for part 1), and postmenopausal subjects age 35-65 years (for part 2)
* Body mass index (BMI) between 18-30 kg/m², inclusive.
* For men: normal values of testosterone (175-781 ng/dL) and LH (1.24-8.62 U/L).
* Women must be postmenopausal for at least 2 years with postmenopausal FSH level according to the local lab (+negative pregnancy test at screening & admission).

Exclusion Criteria:

* smoking
* drug or alcohol abuse
* hypersensitivity to any of the ingredients of the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of GLPG0492 in terms of adverse events, vital signs, ECG and abnormal lab tests in comparison with placebo | Up to 7 to 10 days after last treatment
  Occurrence of adverse events, vital signs, ECG and abnormal lab tests as a measure of safety and tolerability
In male volunteers: effect on protein synthesis in muscle, as measured by the uptake into the muscle of intravenously infused phenylalanine | One week
  During a 5-hour infusion of phenylalanine two muscle biopsies will be taken; this procedure is performed before and after one week of treatment with GLPG0492, to determine the effect of the compound.

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile and metabolism after single and multiple oral doses of GLPG0492 | Up to 24h hours after last treatment
  The plasma levels of GLPG0492 will be determined as a measure of pharmacokinetics, and the plasma and urine samples will be used for metabolism investigation
In female volunteers: effects on hormone household. | up to 7 to 10 days after treatment.
  In female volunteers the effect of two weeks treatment on hormone levels in the blood will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Namour, MSc, Study Director — Galapagos SASU
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium